CLINICAL TRIAL: NCT01416012
Title: Health Related Quality of Life Effects of Off-the-shelf Computer Gaming in Alzheimer and Related Disorders Populations
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 11-PP-06
Record Dates: First submitted 2011-06-30; First posted 2011-08-12 (Estimated); Last update posted 2024-03-18 (Actual); Status verified 2014-06

CONDITIONS: Disease Alzheimer
MeSH Terms: conditions — Alzheimer Disease | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group Kinect (Experimental): Use of the available Kinect games on the Xbox to train balance and gait
  Interventions: Behavioral: Kinect
- Physical Therapy Standard (Active Comparator): This group consists of the usual physical therapy rehabilitation with a special emphasis on lower and upper limb and balance reinforcement.
  Interventions: Behavioral: Physical Therapy (standard)
- Group Nintendo (Experimental): Use of video games available Balance and Gait training in Individualized training sessions.
  Interventions: Behavioral: Balance and Gait training in Individualized sessions
- Group Xbox Kinect (MK) (Experimental): The NW group consists of the use of Nintendo Wii games that targeted upper and lower limbs as well as balance reinforcement
  Interventions: Behavioral: Group Xbox Kinect

INTERVENTIONS:
Behavioral: Physical Therapy (standard) — This group consists of the usual physical therapy rehabilitation with a special emphasis on lower and upper limb and balance reinforcement.
  Arms: Physical Therapy Standard
Behavioral: Balance and Gait training in Individualized sessions — The NW group consists of the use of Nintendo Wii games that targeted upper and lower limbs as well as balance reinforcement.
  Arms: Group Nintendo
Behavioral: Kinect — The NW group consists of the use of Nintendo Wii games that targeted upper and lower limbs as well as balance reinforcement
  Arms: Group Kinect
Behavioral: Group Xbox Kinect — The NW group consists of the use of Nintendo Wii games that targeted upper and lower limbs as well as balance reinforcement
  Arms: Group Xbox Kinect (MK)

SUMMARY:
Interactive games (virtual reality) have recently been the center of interest and scientific discussion in the field of cognitive and functional rehabilitation. From their entertaining and contextual aspects, off-the-shelf video games are potentially interesting tools as adjunct to the patient care, especially for maintaining instrumental activities of daily living (IADL) autonomy.

Disease and physical inactivity worsen the patient's ability in the IADLs, thus reducing health related quality of life (HRQL). This decrease in cognitive and functional abilities can be slowed down using adapted rehabilitation program.

However, there is no randomized controlled study comparing usual physical therapy to virtual reality gaming consoles such as the Nintendo Wii or the Xbox 360 Kinect.

Off-the-shelf gaming consoles offer a large range of games where cognitive and functional abilities from geriatric patients could be stimulated and consequently HRQL improved.

However, a better knowledge of the potential cognitive and functional improvement processes from virtual reality rehabilitation in institutional routine is needed to enhance the quality and the range of the available care in old adults.

This study will not only be a validation platform of virtual reality as stand alone rehabilitation process but also will assess the cost effectiveness of off-the-shelf gaming consoles in HRQL improvement of old adults.

The investigators will compare the efficacy of two off-the-shelf gaming consoles in HRQL changes of patients with Alzheimer disease and related disorders.

•Method

This study is a randomized controlled trial that comprises two study phases :

Phase one; comparing three parallel groups where therapists and assessors will be kept blind of study objectives, and Phase two, the investigators will take the most cost-effective gaming console from phase one (Nintendo Wii or Xbox 360 Kinect) and the investigators will use it as an adjunct to physical therapy compared to physical therapy alone, with respect to the same amount of rehabilitation time.

The interventions are of 120min/week for 6 weeks and a follow-up at 4 weeks after intervention.

Patients will be randomized in either Xbox 360 Kinect group - a Nintendo Wii group - or physical therapy as the 'gold' standard condition.

All groups will receive the same amount of rehabilitation time. Power and sample calculation for phase two will be based on phase one results.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand complex instruction
* Patients with Mild Cognitive Impairment, Alzheimer, Vascular or Alzheimer with cerebro-vascular components dementia.

Geriatric patients with a cognitive level as described by the MMSE between 16 and 26.

* Aged 60 and older
* Signed informed consent (patient or career)

Inclusion criteria for investigator center

* Having a recruitment line from Memory center, outpatient clinic, daycare, nursing homes and long term care
* Able to include 60 patients or more
* Have the French main investigator protocol reviewed and validated by their local ethical committee.

Exclusion Criteria:

* Other type of dementia, psychiatric patients or patients with deemed behavioural disturbances
* Patients using wheelchair for mobility
* Patient with severe deficit in alertness, vision or motor functioning.
* Bedridden patients

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2011-10; Primary Completion 2011-10 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
questionnaires on quality of life | 16 weeks for each test
  * EQ-6D
  * BERG test
  * Timed Up and Go Test and dual task TUG test
  * Engagement using the Observational Assessment of Engagement (OME)

SECONDARY OUTCOMES:
tests on health | 16 weeks for each test
  * Trail making Test A and B
  * Visual Association Test
  * Mini Mental State Examination
  * Neuropsychiatric Inventory
  * Apathy Inventory
  * Strength of lower and upper limbs using dynamometer.
  * Rapid stepping test
  * 10 meters walk test

CONTACTS AND LOCATIONS:
Overall Officials: Robert Philippe, PHD, Principal Investigator — CHU de Nice - CM2R - Hôpital de Cimiez - 4 avenue reine victoria - 06 003 Nice cedex 1
Locations (3):
- The University of Queensland, Saint Lucia, Australia
- CHU de Nice - 4 avenue Reine Victoria - Hôpital de Cimiez, Nice, Alpes-Maritimes, France
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands